CLINICAL TRIAL: NCT00172822
Title: Appendicitis With Medical Treatment
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 940701
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2005-09-15 (Estimated); Status verified 2005-06

CONDITIONS: Appendicitis
Keywords: appendicitis
MeSH Terms: conditions — Appendicitis

STUDY DESIGN:
Observational Model: Natural History | Time Perspective: Prospective

SUMMARY:
prospective study to collect data of patients with appendicitis, not receiving operation

DETAILED DESCRIPTION:
using ultrasound to follow up the resolution of acute appendicitis

ELIGIBILITY:
Inclusion Criteria:patients with appendicitis, not receiving operation -

Exclusion Criteria:nil

-

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80
Dates: Start 2003-01; Study Completion 2005-06

CONTACTS AND LOCATIONS:
Overall Officials: Wan-Ching Lien, MD, Study Director — NTUH
Locations (1):
- Lien, Taipei, Taiwan